CLINICAL TRIAL: NCT00414843
Title: A Prospective Study of Human Bile and Molecular Predictors of Biliary Malignancy Risk
Brief Title: Storage of Bile From Routine Procedures to Study Risk Factors
Status: Terminated | Type: Observational
Why Stopped: Decreasing interest in using samples; department infrastructure waned
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Other Study IDs: 0611-55; IUCRO-0176
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Gallbladder Cancer; Cholangiocarcinoma; Biliary Tract Cancer
Keywords: Storage; Bile; Biomarkers; biliary malignancies
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma; Biliary Tract Neoplasms

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Bile, plasma

SUMMARY:
The purpose of the study is to establish a repository of human bile as a resource for studies evaluating molecular predictors of biliary cancer risk.

DETAILED DESCRIPTION:
The specific aim of this study is to establish a repository of human bile to serve as a resource for studies looking at molecular predictors of biliary tract cancer. The development of fluid based biomarkers will enable early diagnosis in at-risk individuals with a recognized risk factor for cholangiocarcinoma, as well as provide surveillance mechanisms for screening populations where biliary tract cancer has a high incidence.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to IU for treatment of biliary tract disease; Age greater than or equal to 18

Exclusion Criteria:

* Problems other than biliary tract disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to Indiana University for treatment of biliary tract disease.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2006-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Establish Repository of Human Bile | 2024
  Establish a repository of human bile that will serve as a resource through which studies can be performed looking at molecular predictors of biliary tract cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Maluccio, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States